CLINICAL TRIAL: NCT01645982
Title: Comparative Analysis of Cerebral Oximetry and Mean Arterial Pressures at the Cerebral Level in the Beach Chair Position
Status: Completed | Type: Observational
Sponsor: Paul Papagni (Other)
Responsible Party: Sponsor-Investigator, Paul Papagni, Clinical Research Administrator, Holy Cross Hospital, Florida
Organization: Holy Cross Hospital, Florida (Other)
Other Study IDs: 20120943
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2016-02

CONDITIONS: Cerebral Perfusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the changes measured by Somanetics Invos cerebral oximeter to the mean arterial pressure at brain level in patients having elective shoulder replacement surgery. The Somanetics Invos System measures and monitors the oxygen saturation (rS02) of blood in the brain tissues to help prevent brain injury or other complications. The investigators hypothesize that maintaining normocarbia and systemic mean arterial pressure at or above 70mmHg during general anesthesia in the beach chair position will decrease the number of cerebral deoxygenation events during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing elective shoulder replacement surgery
* Subjects must have an ASA class of I or II
* Subject is able and willing to sign the informed consent
* Subject is 18 years of age or older at time of consent
* Subject is not pregnant
* Subject is not a prisoner

Exclusion Criteria:

* Subject has a mental condition that may interfere with the subject's ability to give informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the subject cannot understand the informed consent process, global dementia, prior strokes that interfere with Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject is younger than 18 years of age at consent
* Subject is pregnant
* Subject is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic; Patients undergoing elective shoulder surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Holy Cross Orthopedic Research Institute, Fort Lauderdale, Florida, United States